CLINICAL TRIAL: NCT01542749
Title: Pilot Research Study to Asses Total Body Albumin Levels
Brief Title: Total Body Albumin Measurement Utilizing a Modification of the BVA 100 Blood Volume Analyzer
Status: Completed | Type: Observational
Sponsor: Daxor Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DAXOR 01
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Hypoalbuminemia; Heart Failure; Nephrosis; Cirrhosis; Shock
Keywords: BVA-100 Blood volume analyzer; Human serum albumin labeled with Iodine 131
MeSH Terms: conditions — Hypoalbuminemia; Heart Failure; Nephrosis; Fibrosis; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The DAXOR Corporation manufactures and distributes a blood volume analyzer. The analysis is based on the tracer dilution principle utilizing radioiodine labeled human serum albumin. In addition to calculating human blood volume it is hypothesized that measurement of the dilution of the tracer can also yield an accurate measurement of total body albumin.

DETAILED DESCRIPTION:
Twenty adult individuals underwent a standard blood volume measurement. The specimens for this determination are normally collected over a period of approximately 40 minutes. For the determination of total body albumin, additional specimens were collect over a three to four day period until the counts in the blood specimens were stable. Calculation of the degree of dilution over this time interval is thought to represent dilution of the tracer in albumin in both the intra and extravascular space. The ratio of albumin in the intravascular to the extravascular space is available in the medical literature. The total volume in which the tracer is distributed can be determined from the dilution determined. A calculation of total body albumin is therefore possible. Computation of the total body albumin for the test subjects (all normal individuals) was consistent with values for total body albumin in the literature. The purpose of the development of this method is to permit clinicians to determine albumin status in patients with disturbances in albumin such as burn patients, cirrhotic patients, nephrotic patients as well as patients with protein losing gastroenteropathies.

ELIGIBILITY:
Inclusion Criteria:

* Normal adult males and females.
* Females in the childbearing age group to have test to exclude pregnancy

Exclusion Criteria:

* Children,
* pregnant females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult male and female volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-01; Primary Completion 2010-08 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Total Body Albumin
  The study demonstrated that total body albumin can be determined utilizing modified software designed for this purpose with the BVA 100 blood volume analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Feldschuh, MD, Principal Investigator — Daxor Corporation